CLINICAL TRIAL: NCT00824642
Title: Effect of Acu-TENS on Post-Exercise Expiratory Flow Rate in Subjects With Asthma- A Randomized Controlled Trial
Brief Title: Effect of Acu-Transcutaneous Electrical Nerve Stimulation (TENS) on Post-Exercise Expiratory Flow Rate in Subjects With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice YM Jones, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRE-2004.362
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Asthma
Keywords: Asthma; Exercise training; TENS; Acupuncture; FEV1
MeSH Terms: conditions — Asthma | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group 1 (Experimental): Applied Acu-TENS prior to exercise
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Group 2 (Experimental): Applied Acu-TENS prior to and during exercise
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Group 3 (Placebo Comparator): Applied placebo TENS prior to exercise
  Interventions: Device: placebo

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Applied 45 minutes prior to exercise
  Arms: Group 1; Group 2
Device: placebo — placebo TENS applied prior to exercise
  Arms: Group 3

SUMMARY:
The objective of this study is to investigate the effectiveness of Acu-TENS (Transcutaneous electrical nerve stimulation applied on acupoints) on the post- exercise expiratory flow rate and exercise performance on the subjects with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with asthma attending regular follow up at respiratory clinic

Exclusion Criteria:

* Allergic to gel
* Suffered from other neurological or cardiovascular or musculoskeletal disorders that may affect their exercise performance
* Suffered from upper respiratory tract infection prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) and Forced vital capacity (FVC) | measured before exercise, immediately after exercise and at 20, 40 and 60 minutes post exercise

SECONDARY OUTCOMES:
RPE, Exercise duration | immediately post exercise

CONTACTS AND LOCATIONS:
Overall Officials: Alice Jones, PhD, FACP, Principal Investigator — Department of Rehabilitation Sciences, Hong Kong Polytechnic University
Locations (1):
- Cardiopulmonary and exercise physiology laboratory, The Hong Kong Polytechnic University, Hong Kong, Hong Kong